CLINICAL TRIAL: NCT06386692
Title: Community-based Promotion of Physical Activity in a Semi-urban Area of Pokhara Metropolitan City, Nepal: a Cluster-randomized Controlled Trial
Brief Title: Community Based Promotion of Physical Activity in Nepal (COBIN-PA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Aarhus111
Record Dates: First submitted 2024-04-23; First posted 2024-04-26 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2024-11

CONDITIONS: Exercise
Keywords: Physical activity; Non-communicable disease; Nepal
MeSH Terms: conditions — Motor Activity; Noncommunicable Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PA promotion intervention (Experimental): Behavioral: FCHV visit
  - FCHVs will provide family based physical activity educational intervention through household visit in selected households monthly for 3 months.
  Interventions: Behavioral: FCHVs-led community based educational physical activity intervention
- Wait-list control (No Intervention): No intervention

INTERVENTIONS:
Behavioral: FCHVs-led community based educational physical activity intervention — This intervention will be designed to promote physical activity among adults
  Arms: PA promotion intervention

SUMMARY:
Globally, one in four adults does not meet the WHO-recommended level of physical activity. Insufficient physical activity is the fourth leading risk factor, contributing to 9% of global premature mortality. PA is effective in weight management, cardiorespiratory fitness, and increasing quality of life. However, there is lack of evidence on effectiveness on promoting physical activity in community level. The aim of the study is to test the effectiveness of Female Community Health Volunteers (FCHVs)-led community-based educational program on physical activity promotion in community level. This is an open label cluster-randomized controlled trial with 1:1 allocation where FCHVs will deliver a family-based education for the promotion of physical activity at community level in Nepal. The intervention package will be guided by Theory of planned behavior and will contain home-based interactive health education sessions focused on increasing PA in a household setting. FCHVs will use resource materials for health education. The mixed-effect linear regression model will determine the adjusted interaction between time and intervention. The results of this study will show the changes in the mean moderate to vigorous physical activity minutes per day due to time intervention interaction. The evidence generated from this study will help to provide new knowledge on the community-based promotion of Physical Activity and its effectiveness for policymakers and researchers. It will hopefully support the attainment of the national and global target of reducing insufficient physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 69 years
* without the intention of migrating out of the area for the next 6 months

Exclusion Criteria:

* Those severely ill
* History of mental illness
* Decline to provide consent

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-04-10 (Actual); Study Completion 2025-04-10 (Actual)

PRIMARY OUTCOMES:
Mean moderate to vigorous physical activity | 6 months
  Change in mean moderate-to-vigorous physical activity per day

CONTACTS AND LOCATIONS:
Locations (1):
- Nepal Development Society, Pokhara, Gandaki, Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shrestha R, Adhikari TB, Khatri B, Neupane D, Paudel S, Nielsen RO, Skejo SD, Vaidya A, Kallestrup P. Community-based promotion of physical activity in Nepal: study protocol for a cluster-randomized controlled trial. Trials. 2025 May 24;26(1):170. doi: 10.1186/s13063-025-08885-9. PMID 40413519